CLINICAL TRIAL: NCT02304445
Title: Trans-Arterial Chemo-Embolization (TACE) Vs. TACE Plus Stereotactic Body Radiosurgery (SBRT) in the Treatment of Hepatocellular Carcinoma (HCC)
Brief Title: Chemoembolization With or Without Stereotactic Body Radiosurgery for Liver Cancer
Acronym: TACE-SBRT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Necessary equipment could not be obtained.
Sponsor: Juan Sanabria, MD (Other)
Responsible Party: Sponsor-Investigator, Juan Sanabria, MD, Physician Surgical Oncology, Midwestern Regional Medical Center
Organization: Midwestern Regional Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MZ2014022
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Radiotherapy; Chemoembolization
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transarterial Chemoembolization (TACE) (Active Comparator): Subjects will randomized receive one TACE treatment then receive observation or up to 3 additional TACE treatments as clinically indicated.
  Interventions: Procedure: Transarterial Chemoembolization (TACE)
- TACE+Stereotactic Body Radiotherapy (Experimental): Subjects will receive one TACE treatment then receive 1-5 Stereotactic Body Radiotherapy treatments.
  Interventions: Procedure: Transarterial Chemoembolization (TACE); Radiation: TACE+Stereotactic Body Radiotherapy

INTERVENTIONS:
Procedure: Transarterial Chemoembolization (TACE) — TACE is a treatment modality where local delivery of an anti-neoplastic agent is performed through the feeding artery of the tumor followed by end embolization of the artery. The goal of TACE is to cause tumor necrosis and tumor control via acute arterial occlusion while preserving as much functional liver tissue as possible.
Radiation: TACE+Stereotactic Body Radiotherapy — This intervention adds Stereotactic Body Radiation (SBRT) to TACE therapy. SBRT is the precise administration of large doses of radiotherapy delivered over 1-5 treatments to extra-cranial tumors.
  Arms: TACE+Stereotactic Body Radiotherapy

SUMMARY:
This is a randomized, open-label, active comparator-controlled trial of subjects with advanced (Barcelona stage B/C) hepatocellular carcinoma. Subjects will be receive one treatment with Trans-Arterial Chemo-Embolization (TACE) prior to randomization. Subsequently, subjects will be randomized to observation or, if indicated, up to an additional TACE treatments, or to Stereotactic Body Radiotherapy (SBRT). Tumor response following interventions will be evaluated at three months.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma (Barcelona Stage B or C)
* Treatment with Stereotactic Body Radiosurgery can occur within 6 weeks of enrollment
* Age ≥ 18 years and ≤ 70 years
* Eastern Cooperative Oncology Group Performance status ≤ 2
* Patient has a) Radiographic enhancing liver lesions with early wash out on triple phase CT or MRI or b) histological confirmation of HCC as determined by the Liver Tumor Board
* Hemoglobin > 10.0 g/dL
* Total bilirubin > 3.0 mg/dL
* AST (SGOT) ≤ 3x institutional upper limit of normal
* ALT (SGPT) ≤ 3x institutional upper limit of normal
* Absolute neutrophil count ≥ 1,500/μl
* Platelet count ≥ 50,000/μl (may be post-transfusion if clinically indicated)
* Aggregate maximal dimension of liver tumors ≤ 8 cm
* Cirrhosis classified as Child Pugh Class A or B (score ≤ 7)
* Determined by the treating physician to be medically eligible for liver transplantation measured by imaging modality (MRI/CT scan) three months post final treatment
* Life expectancy ≥ 12 weeks
* Ability to understand study and provide legally effective written informed consent
* Women of child-bearing potential must have a negative test within 4 weeks to the start of the SBRT treatment and must not be pregnant or nursing a child
* Sexually active women must agree to use accepted forms of birth control throughout the study, which include abstinence, oral contraceptives (birth control pills), IUD, diaphragm with spermicide, Norplant, hormone injections, condoms with spermicide, or documentation of medical sterilization

Exclusion Criteria:

* History of abdominal radiation
* Cirrhosis classified as Child Pugh Class B with score ≥ 8
* Prior invasive malignancy other than primary liver malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Evidence of metastatic disease prior to registration
* Evidence of main portal vein thrombosis
* History of cardiac ischemia or stroke within 6 months prior to enrollment
* Any concurrent medical or psychosocial condition that prohibits a major surgical procedure or immunosuppressant that would constitute a contraindication to liver transplantation
* History of sorafenib therapy within 21 days prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | 3 months
  Tumor Response Rate of stage B or C Hepatocellular Carcinoma using TACE vs. TACE plus SBRT at 3 months

SECONDARY OUTCOMES:
Tumor down staging | 3 and 6 months
  Incidence of down staging of stage B or C Hepatocellular Carcinoma using TACE plus SBRT when compared to TACE at 3 and 6 months
Frequency of adverse events | 6 months
  Incidence of Grade 3 or 4 adverse events associated with SBRT for liver tumors
Incidence of local tumor progression | 6 months
  Incidence of local progression as demonstrated by radiological imaging (RECIST criteria)
Number of patients eligibility for liver transplantation | 3 months
  Number of patients achieving sufficient tumor response to attain eligibility for liver transplantation.

OTHER OUTCOMES:
Overall survival | 3 years
  Determination of the number of subjects alive at 3 years following their final study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Sanabria, MD, Principal Investigator — Midwestern Reginal Medical Center